CLINICAL TRIAL: NCT01402908
Title: A Prospective, Randomized, Double-blind, Placebo Controlled, Parallel-group, International Multicenter Phase III Trial of PI-88 in the Adjuvant Treatment of Subjects With Hepatitis Virus Related HCC After Surgical Resection
Brief Title: A Phase III PI-88 in the Adjuvant Treatment of Subjects With Hepatitis Virus Related HCC After Surgical Resection
Acronym: PATRON
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to Interim Analysis and business concerns
Sponsor: Cellxpert Biotechnology Corp. (Industry)
Collaborators: Medigen Biotechnology Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-PI-31
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Results first posted 2020-12-30 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Cancer; Liver Cancer; Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; PI-88; Phase III; Adjuvant Therapy; Hepatoma; Liver Cancer
MeSH Terms: conditions — Neoplasms; Liver Neoplasms; Carcinoma, Hepatocellular | interventions — phosphomannopentaose sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PI-88 (Experimental): Arm 1
  Interventions: Drug: PI-88
- Placebo (Placebo Comparator): Arm 2
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PI-88 — Lyophilized powder reconstituted to provide 160 mg of PI-88
  Other Names: Muparfostat
  Arms: PI-88
Other: Placebo — Lactose lyophilized powder
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if PI-88 is effective and safe in patients who have had surgery to remove primary liver cancer.

DETAILED DESCRIPTION:
Primary liver cancer (hepatocellular carcinoma or HCC) is the fifth most common cancer worldwide. Surgery to remove the tumour remains the principal form of treatment for liver cancer, however recurrence of the disease after surgery is common and survival after recurrence is poor. At the moment there is no recommended standard treatment for HCC immediately after the tumour has been removed surgically. PI-88 is a new experimental drug which blocks the growth of new blood vessels in tumours to stop the tumour growing (starves it of food) and also stops tumour cells spreading. Previous experience with PI-88 has shown it has been well tolerated and has shown some benefit in delaying the time it takes for the hepatocellular carcinoma to reappear after surgery. The purpose of this study is to determine if PI-88 is effective and safe in patients who have had surgery to remove primary liver cancer.

ELIGIBILITY:
Key inclusion criteria:

1. Histologically-proven primary hepatocellular carcinoma with curative resection performed in the 4 - 6 weeks prior to randomization.
2. Age ≥ 18 years.
3. Written, signed and dated informed consent to participate in study
4. ECOG performance status 0 to 1
5. Child Pugh score ≤ 8
6. Platelet count ≥ 80 x 109 cells/liter
7. PT-INR ≤ 1.3
8. aPTT ≤ upper limit of normal

Key exclusion criteria:

1. Pathological confirmation of single tumor < 2 cm in diameter which obtained from the most recent hepatectomy.
2. History of immune-mediated thrombocytopenia other platelet abnormalities or other hereditary or acquired coagulopathies, or laboratory evidence of anti-heparin antibodies, or any previous history of having tested positive for anti-heparin antibodies.
3. Any evidence of tumor metastasis or co-existing malignant disease
4. Any prior recurrence of HCC or any liver resection prior to the most recent procedure
5. Clinically significant non-malignant disease including, but not limited to, surgery within 6 weeks of randomization (apart from liver resection and re-operation for complications of liver resection), active clinically significant infection within 6 weeks prior to randomization, myocardial infarction within 6 months prior to randomization, cerebrovascular event within 12 months prior to randomization or clinically-significant gastrointestinal bleeding within 12 months prior to randomization. Subjects who have experienced post-operative complications of liver resection may be enrolled providing that such complications are fully resolved at the time of screening.
6. Subjects with uncontrolled infection or serious infection within the past 4 weeks.
7. History of prior HCC therapy including chemotherapy, radiotherapy, molecular targeting agents, vaccines, transarterial embolization (TAE), transarterial chemoembolization (TACE), liver transplantation or surgical resection prior to the most recent hepatectomy, at any time prior to randomization. This includes pre-, peri- and post-operative treatments. Pre-operative portal vein embolization is permitted. Subjects should not be enrolled if, at the time of randomization, it is planned that they will subsequently undergo liver transplantation regardless of tumor recurrence.
8. Concomitant use of aspirin (> 150 mg/day), vitamin K antagonists (other than low-dose prophylactic use), heparin within two weeks prior to randomization, or other anti-platelet drugs (e.g. abciximab, clopidogrel, dipyridamole, ticlopidine and tirofiban). Low dose aspirin (≤ 150 mg/day) and low-dose prophylactic vitamin K antagonists (e.g. warfarin ≤ 1 mg/day) are permitted as concomitant medications.
9. History of allergic, anaphylactic or other significant adverse reaction to radiographic contrast media (iodinated or non-iodinated), which cannot be managed by pre-treatment with agents such as steroids or anti-histamines, and which, in the opinion of the investigator, renders the subject unsuitable for routine CT scanning. Subjects who are contra-indicated for CT scanning for other reasons (e.g. ferromagnetic implants, profound claustrophobia), should not be enrolled.
10. Subjects with history of inflammatory bowel disease, any other abnormal bleeding tendency, or subjects at risk of bleeding due to open wounds or planned surgery.
11. Women who are pregnant or breast-feeding or women of child-bearing potential who are unable or unwilling to practice a highly effective means of contraception.
12. Active substance abuse, including alcohol, which, in the opinion of the investigator, risks impairing the ability of the subject to comply with the protocol.
13. Subjects who received other investigational or anti-neoplastic medication within the past 4 weeks.
14. Current participation in any other clinical study or research project which involves administration of a pharmaceutical product or experimental treatment, or which involves protocol-specified laboratory tests, imaging studies or other investigations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2011-08; Primary Completion 2014-07 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Jer Chen, MD, Principal Investigator — National Taiwan University Hospital
Locations (25):
- China (4):
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Peking Union Medical College Hospital, Beijing
  - The General Hospital of People's Liberation Army (301 hospital), Beijing
  - Fudan University Zhongshan Hospital, Shanghai
- Queen Mary Hospital, Hong Kong, Hong Kong
- South Korea (11):
  - Kyungpook National University Hospital (KNUH), Pusan
  - Pusan National University Hospital (PNUH), Pusan
  - Pusan National University Yangsan Hospital (PNUYH), Pusan
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Ajou University Hospital, Suwon
- Taiwan (9):
  - Changhua Christian Hospital, Changhua
  - Chang Gung Memorial Hospital, Kaohsiung City
  - E-Da Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital-Linkou Medical Centre, Taoyuan District

REFERENCES:
- [Derived] Gnoni A, Santini D, Scartozzi M, Russo A, Licchetta A, Palmieri V, Lupo L, Faloppi L, Palasciano G, Memeo V, Angarano G, Brunetti O, Guarini A, Pisconti S, Lorusso V, Silvestris N. Hepatocellular carcinoma treatment over sorafenib: epigenetics, microRNAs and microenvironment. Is there a light at the end of the tunnel? Expert Opin Ther Targets. 2015;19(12):1623-35. doi: 10.1517/14728222.2015.1071354. Epub 2015 Jul 27. PMID 26212068

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PI-88 | Placebo
Started | 258 | 261
Completed | 224 | 243
Not Completed | 34 | 18
Not completed — Withdrawal by Subject | 30 | 17
Not completed — Lost to Follow-up | 3 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT population, defined as all subjects who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | PI-88 | Placebo | Total
Number analyzed (Participants) | 258 | 261 | 519
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.12 (10.201) | 55.08 (9.619) | 54.61 (9.915)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 44 | 96
  Male | 206 | 217 | 423
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Korea | 106 | 96 | 202
  Hong Kong | 6 | 3 | 9
  China | 24 | 24 | 48
  Taiwan | 122 | 138 | 260
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.95 (3.261) | 23.74 (3.015) | 23.84 (3.138)
Liver Cirrhosis (Pre-Operative) [Count of Participants; unit: Participants]
  Missing | 2 | 6 | 8
  None | 105 | 94 | 199
  Mild | 109 | 130 | 239
  Moderate | 35 | 22 | 57
  Severe | 7 | 9 | 16
Total CLIP Score (categorized) [Number; unit: units on a scale] — The Cancer of the Liver Italian Program (CLIP) score is a prognostic staging system for hepatocellular carcinoma.
  It is calculated by assigning a score (0, 1 or 2) to the four clinical factors Child-Pugh stage (0 to 2), tumor morphology (0 to 2), AFP (0 and 1), and portal vein thrombosis (0 and 1). The total score is the sum of the four factors ranging from 0 to 6 and the higher the total score indicates the poorer prognosis.
  units on a scale
    Missing | 1 | 1 | 2
    0 | 146 | 171 | 317
    1 | 83 | 64 | 147
    2 | 19 | 19 | 38
    3 | 7 | 3 | 10
    4 | 2 | 3 | 5
Child-Pugh Stage [Number; unit: units on a scale] — The Pugh-Child score consists of five clinical measures of liver disease including bilirubin, albumin, prothrombin time (or prothrombin time INR), ascites, and encephalopathy. A score of 1, 2, or 3 is given to each measure, with 3 being the most severe. The scores are summed and classified as: class A (well-compensated disease): 5-6 points, class B (significant functional compromise): 7-9 points and class C (decompensated disease): 10-15 points.
  units on a scale
    Missing | 1 | 1 | 2
    A (5 - 6 points) | 256 | 258 | 514
    B (7 - 9 points) | 1 | 2 | 3
Tumor Morphology [Count of Participants; unit: Participants]
  Missing | 1 | 1 | 2
  Uninodular and extension <= 50% | 213 | 228 | 441
  Multinodular and extension <= 50% | 34 | 28 | 62
  Massive or extension > 50% | 10 | 4 | 14
AFP [Count of Participants; unit: Participants] — Blood Alpha-Fetoprotein (APF) level was measured . AFP greater than 400 ng/mL is a sign of hepatoceullar carcinoma. In this report, subjects were grouped into >=400 ng/mL and <400 ng/mL AFP level.
  Participants
    Missing | 1 | 1 | 2
    < 400 ng/ml | 187 | 197 | 384
    >= 400 ng/ml | 70 | 63 | 133
Portal Vein Thrombosis [Count of Participants; unit: Participants]
  Missing | 1 | 1 | 2
  No | 234 | 238 | 472
  Yes | 23 | 22 | 45
ECOG Performance Score [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status scale is used to assess patient's daily living abilities with scores ranging from 0 to 5, and score 0 indicates fully active, where score 5 means dead.
  Participants
    0 | 245 | 247 | 492
    1 | 13 | 14 | 27
Stratification [Count of Participants; unit: Participants] — Subjects were sub-grouped according to vascular invasion and tumor size. V+L+: Vascular Invasion & Tumor Size >= 5 cm V+L-: Vascular Invasion & Tumor Size < 5 cm V-L+: Non Vascular Invasion& Tumor Size >= 5 cm V-L-: Non Vascular Invasion& Tumor Size < 5 cm
  Participants
    V+L+ | 54 | 53 | 107
    V+L- | 70 | 74 | 144
    V-L+ | 33 | 36 | 69
    V-L- | 101 | 98 | 199
Number of Tumors [Count of Participants; unit: Participants]
  1 | 223 | 235 | 458
  2 | 28 | 20 | 48
  >=3 | 7 | 6 | 13
Differentiation of Baseline Tumor [Count of Participants; unit: Participants]
  Missing | 1 | 0 | 1
  Well differentiated | 13 | 20 | 33
  Moderately differentiated | 143 | 117 | 260
  Poorly differentiated | 86 | 103 | 189
  Anaplasia | 15 | 21 | 36
Size of the Largest Explanted Tumor [Count of Participants; unit: Participants]
  <5 cm | 171 | 172 | 343
  5 - <10 cm | 63 | 66 | 129
  >= 10 cm | 24 | 23 | 47
Surgical Margin of Explanted Tumor [Count of Participants; unit: Participants]
  < 10 mm | 118 | 137 | 255
  >= 10 mm | 140 | 123 | 263
  NA | 0 | 1 | 1
Vascular Invasion [Count of Participants; unit: Participants]
  Macro | 18 | 22 | 40
  Micro Only | 106 | 105 | 211
  Absent | 134 | 134 | 268
Baseline Hepatitis Serology [Count of Participants; unit: Participants]
  Missing | 0 | 1 | 1
  HBV+ & HCV+ | 10 | 13 | 23
  HBV+ Only | 212 | 222 | 434
  HCV+ Only | 33 | 20 | 53
  HBV- & HCV- | 3 | 5 | 8
Total Child-Pugh Score (categorized) [Number; unit: units on a scale] — The Pugh-Child score consists of five clinical measures of liver disease including bilirubin, albumin, prothrombin time (or prothrombin time INR), ascites, and encephalopathy. A score of 1, 2, or 3 is given to each measure, with 3 being the most severe. The scores are summed and higher total score indicates worse liver function. The total score ranges from 5 to 15.
  units on a scale
    Missing | 1 | 1 | 2
    5 | 239 | 242 | 481
    6 | 17 | 16 | 33
    7 | 1 | 1 | 2
    8 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Disease-Free Survival (DFS)
Description: To evaluate the efficacy of daily administration of PI-88 versus placebo for the adjuvant treatment of study subjects as measured by DFS during study period.
  As the median DFS could not be estimated, the overall 25 th percentile DFS was reported.
Time Frame: End of study
Population: ITT population, defined as all subjects who were randomized.
Measure: Mean (95% Confidence Interval); unit: weeks
Arm/Group | PI-88 | Placebo
Number analyzed (Participants) | 258 | 261
weeks | 51.0 [28.0 to 52.7] | 75.6 [40.0 to 100.1]

2. Secondary Outcome: Time to Recurrence (TTR)
Description: As no subjects died without a preceding tumor recurrence , no median time to TTR could be estimated in the present study. And therefore the overall 25th percentile DFS was reported.
  The results of time to recurrence (TTR) were the same as that of DFS, as no subjects died without a preceding tumor recurrence.
Time Frame: Time to recurrence (TTR) was defined as the time from randomization to the first time that tumor recurrence was observed or suspected during the study period (3 years).
Population: ITT population
Measure: Mean (95% Confidence Interval); unit: weeks
Arm/Group | PI-88 | Placebo
Number analyzed (Participants) | 258 | 261
weeks | 51.0 [28.0 to 52.7] | 75.6 [40.0 to 100.1]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time, in weeks, from randomization to death from any cause during the study period.
Time Frame: Overall survival was defined as the time, in weeks, from randomization to death from any cause during the study period (3 years).
Population: ITT population
Measure: Mean (Standard Error); unit: weeks
Arm/Group | PI-88 | Placebo
Number analyzed (Participants) | 258 | 261
weeks | 71.7 (0.37) | 69.2 (0.28)

4. Secondary Outcome: Tumor Recurrence Rate (TR Rate)
Description: TR rate was to calculate number of subjects with recurrence among the analyzed population.
Time Frame: The cumulative tumor recurrence rate at weeks 5, 53, 101 and 149 was reported here.
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | PI-88 | Placebo
Number analyzed (Participants) | 258 | 261
Participants
  Cumulative Tumor Recurrence Rate at weeks 5 | 11 | 8
  Cumulative Tumor Recurrence Rate at weeks 53 | 74 | 58
  Cumulative Tumor Recurrence Rate at weeks 101 | 82 | 70
  Cumulative Tumor Recurrence Rate at weeks 149 | 85 | 74

ADVERSE EVENTS:
Time Frame: The adverse events were collected at each study visit during the study period (3 year). In the safety population, the subjects were analyzed according to the actual treatment received and must have received at least one dose of study medication.
Groups:
- PI-88: Arm 1
  PI-88: Lyophilized powder reconstituted to provide 160 mg of PI-88
  In the safety population, the subjects were analyzed according to the actual treatment received and must have received at least one dose of study medication.
  A total of 258 subjects were included in the safety population.
- Placebo: Arm 2
  Placebo: Lactose lyophilized powder
  In the safety population, the subjects were analyzed according to the actual treatment received and must have received at least one dose of study medication.
  Because one subject withdrew the consent before treatment, a total of 260 subjects were included in the safety population.
Arm/Group | PI-88 | Placebo
Serious Adverse Events (participants affected / at risk) | 30/258 | 15/260
Other Adverse Events (participants affected / at risk) | 233/258 | 201/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PI-88 (N=258) | Placebo (N=260)
Cellulitis (Infections and infestations) | 2 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 1 | 0
Mycobacterial infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 1
Injection site cellulitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0
Cervical root pain (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 2 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Branchial cleft cyst (Congenital, familial and genetic disorders) | 0 | 1
Hyperplasia (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PI-88 (N=258) | Placebo (N=260)
Alopecia (Skin and subcutaneous tissue disorders) | 65 | 7
Platelet count decreased (Investigations) | 40 | 13
Injection site haematoma (General disorders) | 34 | 7
Upper respiratory tract infection (Infections and infestations) | 33 | 17
Alanine aminotransferase increased (Investigations) | 32 | 23
Pruritus (Skin and subcutaneous tissue disorders) | 26 | 19
Aspartate aminotransferase increased (Investigations) | 24 | 21
Diarrhoea (Gastrointestinal disorders) | 24 | 13
Rash (Skin and subcutaneous tissue disorders) | 24 | 8
Insomnia (Psychiatric disorders) | 21 | 27
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 21
Neutrophil count decreased (Investigations) | 19 | 3
Injection site haemorrhage (General disorders) | 18 | 0
Abdominal pain upper (Gastrointestinal disorders) | 16 | 12
Alpha 1 foetoprotein increased (Investigations) | 16 | 9
Dizziness (Nervous system disorders) | 16 | 14
Fatigue (General disorders) | 16 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 14
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 | 6
Injection site pain (General disorders) | 13 | 2
Injection site reaction (General disorders) | 13 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No